CLINICAL TRIAL: NCT04793984
Title: Efficacy and Safety Evaluation of Inhaleen Inhalation in Hospitalized COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marinomed Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVID-19/TCP_20_05
Record Dates: First submitted 2021-03-09; First posted 2021-03-11 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Covid19
Keywords: Carragelose; iota-Carrageenan; lung; virus; respiratory virus; inhalation; common cold
MeSH Terms: conditions — COVID-19; Virus Diseases; Respiratory Aspiration; Common Cold

STUDY DESIGN:
Intervention Model Description: randomized placebo-controlled double blinded trial
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaleen (Experimental): Iota-Carrageenan inhalation
  Interventions: Device: Carragelose
- Placebo (Placebo Comparator): NaCl inhalation
  Interventions: Device: NaCl

INTERVENTIONS:
Device: Carragelose — inhalation 3 times a day
  Other Names: iota-Carageenan
  Arms: Inhaleen
Device: NaCl — inhalation 3 times a day
  Other Names: saline
  Arms: Placebo

SUMMARY:
The current study will investigate the tolerability and efficacy of inhaled Carragelose® versus saline in hospitalized COVID-19 patients. As SARS-CoV-2 replicates readily in the lung, it is planed to apply Carragelose® in an inhalative form. Hospitalized COVID-19 patients with respiratory symptoms will inhale Inhaleen for 5 days.

DETAILED DESCRIPTION:
The tolerability and efficacy of inhaled Carragelose® will be investigated in a randomized, double blind, placebo-controlled trial in hospitalized COVID-19 patients.

Patients will inhale Inhaleen or Placebo 3 times a day for 7 minutes for 5 days.

The primary objective of the trial is to demonstrate that Inhaleen inhalation improves the clinical status of hospitalized COVID-19 patients on day 8 compared to placebo inhalation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any trial related procedures are performed
* Age ≥ 18 years
* Hospitalized patients with PCR confirmed SARS-CoV-2 infection and symptom onset ≤ 10 days before randomization
* Patients with respiratory COVID-19 symptoms
* Randomization ≤ 48h from admission
* Peripheral capillary oxygen saturation (SpO2) ≥ 90% on room air or supplemental oxygen at screening
* Patient agrees to refrain from taking other carragelose products (e.g. throat spray, lozenges)

Exclusion Criteria:

* No informed consent
* Persistent hypoxemia with SpO2 < 90% despite supplemental oxygen of > 6LO2/min at screening.
* Patients with predominantly extrapulmonary COVID-19 symptoms (e.g. gastrointestinal, neurological, etc.)
* Subjects who demonstrate respiratory and/or cardiac instability that is considered by the investigator as a reason for exclusion. Additionally, any other clinically significant disease that could interfere with participation in the study, with the intervention being studied, or with the evaluation of symptoms. Specific exclusions are asthma, immune deficiency, autoimmune disease, clinically significant cardiovascular, endocrinological, neurological, respiratory, gastrointestinal disease or any disease that is considered by the investigator as a reason for exclusion.
* Known hypersensitivity or allergy to any component of the test product
* The subject is related to any study personnel or has any other close ties or conflicts of interest with the study sponsor.
* The subject has received any investigational drug or participated in a clinical trial within 4 weeks of entry to this study
* Current medication other than oral contraception,that is considered by the investigator as a reason for exclusion.
* Pregnant/lactating women at the time of recruitment will be excluded from the study
* Participation in another antiviral clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Clinical status of subjects as expressed on the WHO-8-Category ordinal scale: | day 8
  1. Not hospitalized and no limitations of activities
  2. Not hospitalized, with limitations of activities, home oxygen requirement, or both
  3. Hospitalized, not requiring supplemental oxygen and no longer requiring ongoing medical care (used if hospitalization was extended for infections-control or other nonmedical reasons)
  4. Hospitalized not requiring supplemental oxygen but requiring ongoing medical care related to COVID-19) or to other medical conditions)
  5. Hospitalized requiring any supplemental oxygen
  6. Hospitalized requiring non-invasive ventilation or use of high-flow oxygen devices
  7. Hospitalized receiving invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  8. Death

SECONDARY OUTCOMES:
Cycle threshold of SARS-CoV-2 PCR· | until day 15
multiplex viral examination | until day 15
  NxTAG® Respiratory Pathogen Panel + SARS-CoV-2 (Luminex, Cat: X056C0470) detects and differentiates nucleic acids from SARS-CoV-2 and the following organism types and subtypes: Influenza A, Influenza A H1, Influenza A H3, Influenza B, Influenza A 2009 H1N1, Legionella pneumophila, Respiratory Syncytial Virus A, Respiratory Syncytial Virus B, Coronavirus 229E, Coronavirus OC43, Coronavirus NL63, Coronavirus HKU1, Human Metapneumovirus, Rhinovirus/Enterovirus, Adenovirus, Parainfluenza virus 1, Parainfluenza virus 2, Parainfluenza virus 3, Parainfluenza virus 4, Human Bocavirus, Chlamydophila pneumoniae, and Mycoplasma pneumoniae.
supplemental oxygen requirement | until day 15
modified 10 point BORG scale | day 1 to day 5
  a higher score means a worse condition

CONTACTS AND LOCATIONS:
Overall Officials: Arschang Valipour, MD, Principal Investigator — Karl Landsteiner Society; Clinic Floridsdorf; Georg-Christian Funk, MD, Principal Investigator — Karl Landsteiner Society, Clinic Ottakring; Wolfgang Hoeppler, MD, Principal Investigator — Gesundheitsverbund Klinik Favoriten
Locations (1):
- Gesundheitsverbund, Klinik Floridsdorf, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No